CLINICAL TRIAL: NCT01960023
Title: A Phase I/II Dose-Escalation Study Evaluating the Combination of Neratinib and Cetuximab in Patients With "Quadruple Wild-Type" (KRAS/NRAS/BRAF/PIK3CA Wild-Type) Metastatic Colorectal Cancer Resistant to Cetuximab
Brief Title: Safety and Efficacy Study of Neratinib and Cetuximab to Treat Patients With Quadruple Wild-Type Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This registry was planned to report on the Phase II portion of the study. NSABP decided not to proceed with the Phase II portion of the study.
Sponsor: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FC-7
Record Dates: First submitted 2013-09-17; First posted 2013-10-10 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; KRAS; BRAF; NRAS; PIK3CA; NSABP
MeSH Terms: conditions — Colorectal Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — Cetuximab; neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: Cetuximab and Neratinib (Experimental): Cetuximab 400 mg/m2 IV loading dose followed by weekly cetuximab 250 mg/m2 IV plus neratinib per oral daily until disease progression
  Interventions: Drug: Cetuximab; Drug: Neratinib

INTERVENTIONS:
Drug: Cetuximab — 400 mg/m2 IV loading dose followed by weekly cetuximab 250 mg/m2 IV until disease progression
Drug: Neratinib — Phase I portion of the study:
  Dose level 1: 120 mg/day; Dose level 2: 160 mg/day; Dose level 3: 200 mg/day; Dose level 4: 240 mg/day
  Phase II portion of the study: The recommended dose determined in the Phase I portion of the study.

SUMMARY:
The FC-7 study is designed as an open label, single arm, Phase I/II dose-escalation study evaluating the combination of neratinib and cetuximab in patients with metastatic colorectal cancer primary tumor that is "quadruple wild-type " (wild-type KRAS, NRAS, BRAF, PIK3CA). The primary aim in the Phase I portion of this study is to determine the safety and tolerability of the two-drug combination. The primary aim of the Phase II part is to determine the overall objective response rate (complete and partial responses) by Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

Patients will receive concurrent therapy with cetuximab (400 mg/m2 IV loading dose followed by 250 mg/m2 IV weekly), and neratinib.

DETAILED DESCRIPTION:
The neratinib dose-escalation using a 3+3 design will include 4 dose levels (120 mg, 160 mg, 200 mg, and 240 mg) as a daily oral dose. Up to 12 patients will be treated at the maximum tolerated dose (MTD).

The neratinib dose-escalation for the study will proceed on the basis of dose-limiting toxicity (DLT) during cycle 1. DLT will be defined as the occurrence of 1 or more of the following events during cycle 1: any grade diarrhea that is associated with fever or dehydration requiring IV fluids; grade 3 diarrhea lasting more than 2 days on optimal medical therapy; grade 4 diarrhea of any duration; grade 3 or 4 neutropenia associated with fever; grade 4 neutropenia lasting more than 7 days; grade 4 thrombocytopenia; grade 3 or 4 non-hematological toxicity (excluding grade 3 rash or allergic reaction/hypersensitivity); or any toxicity-related delay of more than 2 weeks to initiate cycle 2. Patients will be enrolled at the next dose level when all evaluable patients at the same dose level have completed the first treatment cycle. Enrolled patients will remain on the assigned dose level treatment until toxicity or disease progression.

The Phase II part of this study will proceed with a two-stage design with a maximum of 46 patients. Between 6 and 12 patients at the Phase I MTD level will be included in the Phase II, stage-one analysis.

Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0.

Submission of tumor and blood samples for FC-7 correlative science studies will be a study requirement for all patients. A core biopsy procedure to procure fresh tumor samples from an accessible site of metastasis will be performed before study dose level assignment (after the patient has signed the consent form and has been screened for eligibility).

Optional biopsy samples of metastatic disease will be procured from consenting patients after Cycle 1 of treatment and at the time of disease progression.

ELIGIBILITY:
Inclusion criteria:

* Patients with resected primary must be active participants of the NSABP Patient Registry and Biospecimen Profiling Repository (MPR-1) study. Patients with intact primary and metastatic KRAS wild-type disease at presentation (treatment naive), must have signed consent for quadruple wild-type central testing for treatment-naive tumor sample submission
* The Eastern Cooperative Oncology Group (ECOG) performance status must be 0, 1, or 2.
* Patients must have the ability to swallow oral medication.
* The tumor tissue must have been determined to be KRAS, NRAS, BRAF, PIK3CA wild-type by central CLIA testing.
* There must be documentation by PET/CT scan, CT scan, or MRI, that the patient has evidence of measurable metastatic disease per RECIST criteria.
* Patients must have an accessible metastatic lesion for pretreatment core biopsy procurement.
* Unless either drug is medically contraindicated, patients must have received oxaliplatin and irinotecan as part of standard chemotherapy regimens. (This includes adjuvant therapy.)
* Patients must have had at least one prior treatment for metastatic disease with standard chemotherapy and cetuximab in combination or as monotherapy. [Note: patients who received panitumumab instead of cetuximab are eligible.]
* At the time of study entry, blood counts performed within 4 weeks prior to study entry must meet the following criteria: absolute neutrophil count (ANC) must be greater than or equal to 1000/mm3; Platelet count must be greater than or equal to 100,000/mm3; Hemoglobin must be greater than or equal to 9 g/dL
* The following criteria for evidence of adequate hepatic function performed within 4 weeks prior to study entry must be met: Total bilirubin must be less than or equal to 1.5 x upper limit of normal (ULN); aspartate aminotransferase (AST) and ALT must be less than or equal to 2.5 x ULN for the lab or less than or equal to 5 x ULN if liver metastasis;
* Serum creatinine performed within 4 weeks prior to study entry must be less than or equal to 1.5 x ULN for the lab.
* Female patients and male patients with female partners of reproductive potential must agree to use an effective method of contraception during therapy and for at least 6 months after the last dose of study therapy.
* Patients with acquired immunodeficiency syndrome (AIDS-related illnesses) or known human immunodeficiency virus (HIV) disease must: Have a CD4 count greater than or equal to 200 cells/uL within 30 days prior to beginning study therapy; Be off all antiretroviral therapy (prophylaxis/treatment) greater than 60 days prior to beginning study therapy; Have no evidence of opportunistic infections.

Exclusion criteria:

* Diagnosis of anal or small bowel carcinoma.
* Colorectal cancer other than adenocarcinoma, e.g., sarcoma, lymphoma, carcinoid.
* Previous therapy with any HER2 TKI (such as trastuzumab, lapatinib, neratinib, etc.) for any malignancy.
* Symptomatic brain metastases or brain metastases requiring chronic steroids to control symptoms.
* Active hepatitis B or hepatitis C with abnormal liver function tests.
* Malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease or condition significantly affecting gastrointestinal function.
* Persistent Common Toxicity Criteria for Adverse Effects (CTCAE v4.0) greater than or equal to grade 2 diarrhea regardless of etiology.
* Chronic daily treatment with corticosteroids with a dose of greater than or equal to 10 mg/day methylprednisolone equivalent (excluding inhaled steroids).
* CTCAE v4.0 grade 3 or 4 anorexia or nausea related to metastatic disease.
* CTCAE v4.0 greater than or equal to grade 2 vomiting related to metastatic disease.
* Any of the following cardiac conditions: Documented congestive heart failure; Myocardial infarction within 6 months prior to study entry; Unstable angina within 6 months prior to study entry; Symptomatic arrhythmia
* Serious or non-healing wound, skin ulcer, or bone fracture.
* History of bleeding diathesis or coagulopathy. (Patients on stable anticoagulant therapy are eligible.)
* Symptomatic interstitial lung disease or definitive evidence of interstitial lung disease described on CT scan, MRI, or chest x-ray in asymptomatic patients; dyspnea at rest requiring current continuous oxygen therapy.
* Other malignancies unless the patient is considered to be disease-free and has completed therapy for the malignancy greater than or equal to 12 months prior to study entry. Patients with the following cancers are eligible if diagnosed and treated within the past 12 months: carcinoma in situ of the cervix, colorectal carcinoma in situ, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Previous serious hypersensitivity reaction to monoclonal antibodies. (Determination of "serious" hypersensitivity reaction is at the investigator's discretion.)
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
* Pregnancy or lactation at the time of study entry.
* Use of any investigational agent within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07-13 (Actual); Study Completion 2016-07-13 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of cetuximab and neratinib during the Phase I portion of the study. | From start of study therapy weekly through disease progression or end of therapy, approximately 2 years
  Number of patients experiencing dose limiting toxicities (DLT).
Number of patients with Overall response rate (ORR)(complete response/partial response) and progression free survival (PFS) during the Phase II portion of the study | From start of study through 16 weeks.
  Response as measured by RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS). The time to progression and the time to progression based on tumor HER2 status. | From start of study through disease progression or end of therapy, approximately 2 years
Tumor measurement to determine objective tumor decrease and stable disease | From start of study through desease progression or end of therapy, approximately 2 years
  Measurement of disease status by continuous tumor measurement.
Measure molecular and genetic correlatives for neratinib and cetuximab | Baseline (prior to treatment assignment), prior to therapy, after completion of cycle 1, and at disease progression approximately 2 years.
The frequency and severity of adverse events to evaluate the overall toxicity in the Phase II portion of the study. | From start of study therapy through 30 days after end of therapy, approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (12):
- United States (12):
  - University of Florida, Gainesville, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Decatur Memorial Hospital, Decatur, Illinois
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania

REFERENCES:
- [Derived] Jacobs SA, Lee JJ, George TJ, Wade JL 3rd, Stella PJ, Wang D, Sama AR, Piette F, Pogue-Geile KL, Kim RS, Gavin PG, Lipchik C, Feng H, Wang Y, Finnigan M, Kiesel BF, Beumer JH, Wolmark N, Lucas PC, Allegra CJ, Srinivasan A. Neratinib-Plus-Cetuximab in Quadruple-WT (KRAS, NRAS, BRAF, PIK3CA) Metastatic Colorectal Cancer Resistant to Cetuximab or Panitumumab: NSABP FC-7, A Phase Ib Study. Clin Cancer Res. 2021 Mar 15;27(6):1612-1622. doi: 10.1158/1078-0432.CCR-20-1831. Epub 2020 Nov 17. PMID 33203645